CLINICAL TRIAL: NCT06574139
Title: Evaluation of Unstained
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Policy & Research Group (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Mathematica Policy Research, Inc. (Other); Reproductive Health National Training Center (Unknown); PCI Media (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1 TP2AH000085-01-00
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Teen Pregnancy Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unstained (Experimental)
  Interventions: Behavioral: Unstained
- Like (Sham Comparator)
  Interventions: Behavioral: Like

INTERVENTIONS:
Behavioral: Unstained — Unstained is an individual-level, virtual intervention that involves three ~60-minute sessions delivered over a 3-6 week period. Each session includes watching two videos (six videos total), followed by a discussion facilitated by study coordinators.
  Arms: Unstained
Behavioral: Like — Like is an hour-long film that discusses the impact of social media on the brain. Participants will receive a link to the film and will be asked to watch it independently. The film does not include information related to the outcomes of interest for the study.
  Arms: Like

SUMMARY:
The goal of this randomized trial is to learn if the Unstained intervention has a positive impact on the sexual health behaviors of sexually active youth between the ages of 14 and 22 years old who are at risk for or involved in the legal system. The primary research questions it aims to answer are:

* Three months after being offered the intervention, does Unstained impact youth's receipt of sexually transmitted infection testing in the past four months?
* Nine months after being offered the intervention, does Unstained impact youth's frequency of having vaginal and anal sex without condoms in the past four months?

Researchers will compare participants randomized to receive Unstained (treatment group) to participants randomized to receive a control condition that contains no sexual or reproductive health information (control group).

Participants randomized to the treatment group will be offered Unstained as a virtual, individual-based intervention delivered during three ~60 minute sessions over a 3-6 week period. Participants randomized to the control group will be offered a virtually delivered control condition.

DETAILED DESCRIPTION:
This is an individual-level, randomized control trial to rigorously evaluate the impact of the Unstained intervention. Participant outcomes will be assessed using self-reported, individual-level data gathered using a structured questionnaire administered at three time points: baseline (enrollment); three months post-intervention (five months after baseline); and nine months post-intervention (eleven months after baseline).

ELIGIBILITY:
Inclusion Criteria:

* United States resident
* Owns or has regular access to a personal device with internet access
* Comfortable reading, speaking, and writing in English
* Has had vaginal or anal sex in the past 3 months
* At risk for or involved in the legal system

Exclusion Criteria:

* Currently trying to start a pregnancy
* Currently in jail or being detained in a facility
* Enrolled in an ongoing PRG-run TPP study
* Identified as fraudulent
* Participating in another known OPA-funded research study

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-09-14 (Estimated)

PRIMARY OUTCOMES:
Receipt of sexually transmitted infection (STI) testing in the past four months | Assessed three months after the intervention period has ended (five months post-baseline)
  Participants are asked the following item:
  1) Have you been tested for sexually transmitted infections (STIs) in the past 4 months? The resulting variable is dichotomous with values 0 or 1, where 0 indicates a person who has not received STI testing in the past four months and 1 indicates a person who has received STI testing in the past four months.
Times having vaginal and anal sex without condoms in the past four months | Assessed nine months after the intervention period has ended (11 months post-baseline)
  Participants are asked the following two items:
  1. In the past 4 months, how many times have you had vaginal sex without you or your sexual partner using a condom?
  2. In the past 4 months, how many times have you had anal sex without you or your sexual partner using a condom? The resulting variable is continuous with values that range from 0 to k, where 0 indicates that a person has not engaged in vaginal and anal sex without a condom in the past four months, and k indicates the number of times the person has engaged in vaginal and anal sex without a condom in the past four months.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Walsh, PhD, Principal Investigator — The Policy & Research Group
Locations (1):
- The Policy & Research Group, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
A dataset will be prepared at the conclusion of the study, which includes de-identified individual-level data on all study participants who contributed self-report data. Respondents will be represented only by a research ID number. Included in the dataset will be self-report data collected across all survey administrations (including demographic characteristics, sexual behaviors, and theoretical antecedents to those behaviors) and select information on program participation (e.g., which program components were completed). Basic data cleaning steps will be taken in order to ensure data are unidentifiable and to increase usability.
Supporting Information: SAP
Time Frame: The individual participant dataset will become available twelve months after the study has concluded.